CLINICAL TRIAL: NCT05014841
Title: The Neural Coding of Speech Across Human Languages
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: University of California, Berkeley (Other); Lawrence Livermore National Laboratory (Other); The University of Hong Kong (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: U01NS117765 (NIH); U01NS117765 (NIH)
Record Dates: First submitted 2021-08-13; First posted 2021-08-20 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Epilepsy; Brain Tumor; Speech; Bilingualism
MeSH Terms: conditions — Epilepsy; Brain Neoplasms; Speech

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Electrocorticography (ECoG) recording during Speech Tasks (Experimental): Participants listened to 20-minute Speech Tasks while ECoG signals for neural activity was recorded during their intraoperative procedure or inpatient hospitalization at the University of California, San Francisco (UCSF).
  Interventions: Behavioral: Speech Tasks

INTERVENTIONS:
Behavioral: Speech Tasks — Listen to 20-minutes of speech sounds in English, Spanish, and/or Mandarin.

SUMMARY:
The overall goal of this study is to reveal the fundamental neural mechanisms that underlie comprehension across human spoken languages. An understanding of how speech is coded in the brain has significant implications for the development of new diagnostic and rehabilitative strategies for language disorders (e.g. aphasia, dyslexia, autism, et alia). The basic mechanisms underlying comprehension of spoken language are unknown. Researchers are only beginning to understand how the human brain extracts the most fundamental linguistic elements (consonants and vowels) from a complex and highly variable acoustic signal. Traditional theories have posited a 'universal' phonetic inventory shared by all humans, but this has been challenged by other newer theories that each language has its own unique and specialized code. An investigation of the cortical representation of speech sounds across languages can likely shed light on this fundamental question. Previous research has implicated the superior temporal cortex in the processing of speech sounds. Most of this work has been entirely carried out in English. The recording of neural activity directly from the cortical surface from individuals with different language experience is a promising approach since it can provide both high spatial and temporal resolution. This study will examine the mechanisms of phonetic encoding, by utilizing neurophysiological recordings obtained during neurosurgical procedures. High-density electrode arrays, advanced signal processing, and direct electrocortical stimulation will be utilized to unravel both local and population encoding of speech sounds in the lateral temporal cortex. This study will also examine the neural encoding of speech in patients who are monolingual and bilingual in Mandarin, Spanish, and English, the most common spoken languages worldwide, and feature important contrastive differences of pitch, formant, and temporal envelope. A cross-linguistic approach is critical for a true understanding of language, while also striving to achieve a broader approach of diversity and inclusion in neuroscience of language.

DETAILED DESCRIPTION:
Experimental approaches with significantly greater spatial and temporal resolution are necessary to directly resolve, both local- and population- level, the contrastive encoding of speech sounds. This study proposes an innovative methodological approach using customized intracranial high-density electrode arrays to record neural activity directly from nonprimary auditory cortex in patients undergoing clinical neurosurgical procedures (acute intraoperative and chronic extraoperative). This approach overcomes obstacles in traditional neuroimaging by offering high signal-to-noise recordings, unprecedented detailed spatiotemporal resolution, and a large number of simultaneously recorded cortical sites in awake, behaving subjects. The research study team will leverage the diversity of languages spoken by patients that are treated at the large volume epilepsy and tumor brain mapping programs at the University of California, San Francisco. They will examine cortical responses to speech stimuli (natural speech corpora and control tokens) in Spanish, Mandarin, and English speakers (monolingual and bilingual). They will also focus on encoding models in three fundamental domains of acoustic-phonetic cues that are present in all languages: pitch, formants, and amplitude envelope. The aims of this study seeks to determine how pitch cues encode lexical tone processing in Mandarin (Aim 1), the cortical representation of vowels in Spanish and English (Aim 2), and the encoding of the speech amplitude envelope in Spanish and English (Aim 3). Together, these aims will elucidate mechanistic principles of speech encoding in the human auditory cortex to understand what is shared and different across human spoken languages. Abnormalities in these fundamental processes have been implicated in a host of communication disorders such as dyslexia, developmental language disorder, central hearing loss, and aphasia. These results should heavily impact current theories of speech processing and, therefore, will have significant implications for understanding and remediating human disorders across different languages.

ELIGIBILITY:
Inclusion Criteria:

* Participants with epilepsy or brain tumors at UCSF undergoing surgical electrode implantation for seizure localization or for speech and language mapping and
* Participants with electrodes implanted in at least two regions of interest who are willing and able to cooperate with study tasks.

Exclusion Criteria:

* Participants who lack capacity or decline to provide informed consent,
* Participants who have significant cerebral lesions or
* Participants with cognitive deficits that preclude reliable completion of study tasks.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2015-09-14 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Electrocorticography (ECoG) Signals for Neural Activity Identified During Intraoperative Procedure or Inpatient Hospitalization | Between 10-30 minutes
  Number of participants with ECoG signals for neural activity identified during intraoperative procedure or inpatient hospitalization, between 10-30 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Edward F Chang, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
No Individual Participant Data (IPD) will be made available to other researchers; only de-identified data will be shared with Collaborators for research analysis.